CLINICAL TRIAL: NCT05787886
Title: Clinical Outcomes of Percutaneous Coronary Intervention With Rotational Atherectomy: the Poland Single RA-BIA Registry
Brief Title: Rotational Atherectomy: Long-term Results From a Single Center Experience
Acronym: RA-BIA
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Principal Investigator, Lukasz Kuzma, Assistant Professor, Medical University of Bialystok
Other Study IDs: UMB-KKI-105
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Ischemic Heart Disease; Acute Coronary Syndrome
Keywords: rotational atherectomy; rotablation
MeSH Terms: conditions — Myocardial Ischemia; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The RA-BIA Registry is a single-center observational study. The study included consecutive patients from 2008 who met inclusion criteria and were treated with RA. The main aim of the study is to assess the efficacy of rotational atherectomy.

DETAILED DESCRIPTION:
Severe coronary artery calcifications occur in about 10% of patients undergoing percutaneous coronary intervention (PCI). They constitute a strong independent predictor of an adverse cardiovascular event. Even though the risk factors and pathomechanisms leading to severe coronary calcification are well understood, the options for effective treatment remain insufficient.

In the presence of severe calcification, standard PCI has inferior immediate and long-term outcomes. In this situation, advanced lesion modification techniques are indispensable to improve PCI outcomes. Dedicated balloons and essentially ablative techniques are available. Rotational atherectomy (RA) is the oldest and best-recognized ablative technique. It is generally acknowledged that superficial modification of calcified atherosclerotic lesions is an optimal mechanism of action in RA.

The RA-BIA Registry is a single-center observational study. The study included consecutive patients from 2008 who met inclusion criteria and were treated with RA. The main aim of the study is to assess the efficacy of rotational atherectomy.

The primary endpoints were device-oriented composite endpoint (DOCE) (defined as a composite of cardiac death, TLR, and target vessel MI), TVR, MI, and cardiac death. TVR and TLR were defined according to the definitions of endpoints for clinical trials. The secondary endpoints were the clinical success rate of the RA procedure (defined as successful revascularization of all treated lesions and the incidence of in-hospital complications including coronary perforation, coronary dissection, coronary low flow or no flow, emergency CABG, tamponade, MI, stroke or transient ischemic attack (TIA), bleeding events (according to the Bleeding Academic Research Consortium [BARC] classification and death.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years old
2. Lesions in target vessels requiring RA
3. Patient accepting the appropriate follow-up as per study definition

Exclusion Criteria:

1. Patient age < 18 years
2. Patients who previously participated in this study.
3. Pregnant and/or breastfeeding females or females who intend to become pregnant.
4. Unable to tolerate dual antiplatelet therapy (i.e., aspirin, and either clopidogrel, prasugrel, or ticagrelor) .
5. The subject has an allergy to imaging contrast media which cannot be adequately pre-medicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease who were treated with rotational atherectomy.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2007-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of various endpoints | 5 years
  1. Rate of the device-oriented composite end point (DOCE) defined as a composite of cardiac death, target Lesion Revascularization (TLR), and target vessel MI), Target Vessel Revascularization (TVR), myocardial infraction (MI), and cardiac death.

SECONDARY OUTCOMES:
Procedural, Technical and Clinical Success | 5 years
  1. Procedural Success Defined as successful use of rotational atherectomy
  2. Technical Success Defined as a successful rotational atherectomy with stent implantation
  3. Clinical Success Defined as successful revascularization of all treated lesions and the incidence of in-hospital complications including coronary perforation, coronary dissection, coronary low flow or no flow, emergency CABG, tamponade, MI, stroke or transient ischaemic attack (TIA), bleeding events (according to the Bleeding Academic Research Consortium [BARC] classification and death.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Invasive Cardiology, Medical University of Bialystok, The Medical University of Bialystok Clinical Hospital, Bialystok, Poland